CLINICAL TRIAL: NCT02538146
Title: Acetyl-L-carnitine as Pain Therapy in Chronic Pancreatitis
Brief Title: Effect of Acetyl-L-carnitine on Chronic Pancreatitis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Older participants could not tolerate the acidity of the product and withdrew.
Sponsor: Karin High (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Karin High, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UKentucky
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Chronic Pancreatitis
Keywords: pain; depression; cytokines; well-being
MeSH Terms: conditions — Pancreatitis, Chronic; Pain; Depression | interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Acetyl-L-carnitine 1000mg 2X per day for 3 months
  Interventions: Dietary Supplement: acetyl-L-carnitine 1000mg 2X per day for 3 months

INTERVENTIONS:
Dietary Supplement: acetyl-L-carnitine 1000mg 2X per day for 3 months — non-essential dietary amino acid
  Other Names: ALC

SUMMARY:
An open label pilot study will determine the effect of the amino acid nutritional supplement acetyl-L-carnitine (ALC) on pain, quality of life, well-being, and serum pro-inflammatory mediator and oxidative stress levels in volunteers with chronic pancreatitis. The ALC is given to all participants for 3 months, and assessments will occur at intake and after 3 months.

DETAILED DESCRIPTION:
This is an open label pilot study to determine the effect of the amino acid nutritional supplement acetyl-L-carnitine (ALC) on chronic pancreatitis. ALC is an acetylated form of naturally occurring amino acid L-carnitine ((R)-3-Acetyloxy-4-trimethylammonio-butanoate) found in red meat and is readily commercially available. Supplementation with ALC may decrease pain and improve overall health based on our preclinical treatment studies in rats with high fat and alcohol induced pancreatitis. In rats, ALC reduces pain measures, improves glucose tolerance, decreases lipid peroxidation, and Ki67 cellular injury biomarker, and improves pancreatic histopathology. The measurable outcomes of this clinical study are patients' questionnaire scores for:

pain, quality of life, well-being, and serum pro-inflammatory mediator and oxidative stress levels in volunteers with chronic pancreatitis. The questionnaires are given at intake and at experiment end (3 months). Participants will receive ALC for 3 months. These findings will indirectly determine the effect of ALC on the function and inflammatory state of the pancreas. Currently, there is no specific therapy for chronic pancreatitis, and its pathophysiology is still poorly understood. It is known that chronic pancreatitis is caused by ongoing inflammation in the pancreas, yet, no pharmacological intervention exists that optimally addresses this. The broad actions of ALC as an antioxidant and anti-inflammatory agent as well as its ability to reduce side-effects of alcohol cessation make it a perfect compound to pursue for the treatment of pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with chronic pancreatitis are included.

Exclusion Criteria:

* Patients with pancreatic pseudocysts, abscesses, pseudoaneurysms, pancreatitic fistulas, pancreatic adenocarcinoma,
* Females that are pregnant or lactating
* Children are excluded.
* Patients suffering from seizure or thyroid disorders are also excluded due to possible exaggeration of their symptoms from taking ALC according to manufacturer.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pain score | 3 months
  McGill short form Visual Analogue Scale (VAS scale) 1 normal 2-10 pain level

SECONDARY OUTCOMES:
Well Being | 3 months
  Normal: 0 of 30 days with major impairment; 30 of 30 days feeling very healthy and full of energy
Generalized anxiety disorder 7-item (GAD-7) Scoring | 3 months
  5-< 10 Mild Anxiety 10-<15 Moderate Anxiety >15 Severe Anxiety 5-< 10 Mild Anxiety 10-<15 Moderate Anxiety >15 Severe Anxiety 5-< 10 Mild Anxiety 10-<15 Moderate Anxiety >15 Severe Anxiety 5-< 10 Mild Anxiety; 10-<15 Moderate Anxiety; >15 Severe Anxiety
Patient Depression Questionnaire Scoring | 3 months
  5-<10 Mild Depression; 10-<15 Moderate Depression; 15-<20 Moderately Severe Depression; >20 Severe Depression
Inflammatory Markers | 3 months
  TBARS: in fasted (8 hrs) 4.7±0.2 μmol/l blood serum; TGFbeta1: 20-50 pg/ml; PDGF: 20-30 pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Karin W High, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Center for Clinical and Translational Science, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
One young participant (>35) successfully completed the trial and provided a personal statement and data indicating the acetyl-L-carnatine had improved his pancreatitis. Two older individuals (>60) withdrew from the study within two months citing inability to tolerate the acidity of the product. Difficulties recruiting in this very ill population was also a consideration in termination. For additional information contact sabrina.mcilwrath@uky.edu